CLINICAL TRIAL: NCT06549140
Title: Effects of an Augmented Reality Exercise Program in Older Adults Physical Fitness and Cognitive Abilities
Brief Title: Effects of an Augmented Reality Exercise Program in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Collaborators: Élvio Rúbio Gouveia (Unknown); Hildegardo Noronha (Unknown); Francisco Santos (Unknown); Mara Dionísio (Unknown); Eva Freitas (Unknown); Pedro Campos (Unknown); Paulo Bala (Unknown)
Responsible Party: Principal Investigator, Cíntia Franca, Dr. Cíntia França, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGAMESPRR
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Augmented Reality Exercise Program; Traditional Exercise Program; Control Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Participants were not enrolled in organized exercise programs during the study (12 weeks).
- Traditional exercise program (Experimental): Participants enrolled in a traditional organized exercise program (group sessions) based on two weekly sessions of 45 to 60 minutes each for 12 weeks. These sessions are supervised by sports and exercise professionals, targeting physical fitness components (cardiorespiratory capacity, strength, balance, agility, and flexibility) and cognitive function (reaction time and decision-making).
  Interventions: Other: Traditional exercise program
- Augmented reality exercise program (Experimental): Participants enrolled in an organized exercise program based on two weekly sessions of 45 to 60 minutes each for 12 weeks: one traditional session (group session) and one augmented reality (AR) session (individual session), both supervised by sports and exercise professionals. The AR session was designed to provide a full exercise session targeting physical fitness components (cardiorespiratory capacity, strength, balance, agility, and flexibility) and cognitive function (reaction time, decision-making, and memory).
  Interventions: Other: Augmented reality exercise program

INTERVENTIONS:
Other: Augmented reality exercise program — Participants enrolled in an organized exercise program based on two weekly sessions of 45 to 60 minutes each for 12 weeks: one traditional session (group session) and one augmented reality (AR) session (individual session), both supervised by sports and exercise professionals. The AR session was designed to provide an entire exercise session targeting physical fitness components (cardiorespiratory capacity, strength, balance, agility, and flexibility) and cognitive function (reaction time, decision-making, and memory).
  Arms: Augmented reality exercise program
Other: Traditional exercise program — Participants enrolled in a traditional organized exercise program (group sessions) based on two weekly sessions of 45 to 60 minutes each for 12 weeks. These sessions are supervised by sports and exercise professionals, targeting physical fitness components (cardiorespiratory capacity, strength, balance, agility, and flexibility) and cognitive function (reaction time and decision-making).
  Arms: Traditional exercise program

SUMMARY:
This research aims to examine the effects of an augmented reality (AR) exercise program on physical fitness (cardiorespiratory capacity, strength, balance, agility, and flexibility) and cognitive function (reaction time, decision-making, and memory).

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders
* 60 years or older
* Autonomous community-dwelling older adults

Exclusion Criteria:

* Neurological disorders
* Cognitive impairment
* Health limitations related to exercise participation

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Physical fitness | Testing sessions will occur at baseline, at week 6, at week 13 and at week 18.
  Physical fitness will be assessed using the fitness test battery proposed by Rikli & Jones (1999), including: 30-s chair stand test to assess lower-body strength, arm curl test to evaluate upper-body strength, back scratch test to examine upper-body flexibility, chair seat and reach test to assess lower-body flexibility, 8-foot up-and-go test to assess agility and dynamic balance, and the 6-min walk test to evaluate aerobic endurance.
Physical activity | Participants enrolled in exercise programs will be monitored using accelerometry. Individual data will be collected in all exercise sessions (total of 48 sessions).
  Physical activity levels will be measured using accelerometry during each exercise session.
Body composition | Testing sessions will occur at baseline, at week 6, at week 13 and at week 18.
  Body composition will be evaluated using the InBody 770, which allows a hand-to-foot biolectrical analysis. Bodyweight, body fat percentage, and fat-free mass will be used for analysis.
Cognitive function | The assessment will be conducted at baseline, at week 6, at week 13 and at week 18.
  Participants' cognitive function will be examined through the Cognitive Telephone Screening Instrument and the Mini Mental State Examination.

SECONDARY OUTCOMES:
SF-36 questionnaire | The assessment will be conducted at baseline and at week 13 after the intervention end.
  The SF-36 questionnaire is used to assess the participant's health status of participants. It consists of 36 items that assess physical functioning, physical performance, physical pain, emotional functioning, vitality, mental health, social functioning, and general health. The higher the score, the better the participant's health.

CONTACTS AND LOCATIONS:
Overall Officials: Élvio Gouveia, PhD, Study Director — University of Madeira